CLINICAL TRIAL: NCT02536209
Title: A Study to Investigate the Pharmacodynamic Effect of Single Doses of MT-8554 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MT-8554-E03
Record Dates: First submitted 2015-08-16; First posted 2015-08-31 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Regimen 1 (Experimental): Period 1: MT-8554 low dose, Period 2: MT-8554 high dose, Period 3: Placebo and Period 4: Oxycodone hydrochloride, respectively single dosing
  Interventions: Drug: MT-8554 low dose; Drug: MT-8554 high dose; Drug: Oxycodone hydrochloride; Drug: Placebo
- Regimen 2 (Experimental): Period 1: MT-8554 high dose, Period 2: Oxycodone hydrochloride, Period 3: MT-8554 low dose and Period 4: Placebo, respectively single dosing
  Interventions: Drug: MT-8554 low dose; Drug: MT-8554 high dose; Drug: Oxycodone hydrochloride; Drug: Placebo
- Regimen 3 (Experimental): Period 1: Placebo, Period 2: MT-8554 low dose, Period 3: Oxycodone hydrochloride and Period 4: MT-8554 high dose, respectively single dosing
  Interventions: Drug: MT-8554 low dose; Drug: MT-8554 high dose; Drug: Oxycodone hydrochloride; Drug: Placebo
- Regimen 4 (Experimental): Period 1: Oxycodone hydrochloride, Period 2: Placebo, Period 3: MT-8554 high dose and Period 4: MT-8554 low dose, respectively single dosing
  Interventions: Drug: MT-8554 low dose; Drug: MT-8554 high dose; Drug: Oxycodone hydrochloride; Drug: Placebo

INTERVENTIONS:
Drug: MT-8554 low dose
Drug: MT-8554 high dose
Drug: Oxycodone hydrochloride
Drug: Placebo

SUMMARY:
The purpose of this study is to investigate the pharmacodynamic effect of single doses of MT-8554 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and free from clinically significant illness or disease
* Male Caucasian subjects aged 18 to 55
* A body weight of ≥60 kg

Exclusion Criteria:

* Participation in more than three clinical studies involving administration of an Investigational Medicinal Product (IMP) in the previous year, or any study within 12 weeks.
* Clinically significant endocrine, thyroid, hepatic, respiratory, gastro-intestinal, renal, cardiovascular disease, or history of any significant psychiatric/psychotic illness disorder.
* Clinically relevant abnormal medical history, physical findings or laboratory values

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic effect as measured by Visual Analogue Scale for Cold Pressor Test | up to 10 hours post dosing

SECONDARY OUTCOMES:
Safety and Tolerability as measured by vital signs | up to Day6 of treatment period 4
Safety and Tolerability as measured by ECG | up to Day6 of treatment period 4
Safety and Tolerability as measured by laboratory safety assessments | up to Day6 of treatment period 4
Safety and Tolerability as measured by physical examination | up to Day6 of treatment period 4
Safety and Tolerability as measured by number of participants with adverse events | up to Day6 of treatment period 4
Plasma concentration of MT-8554 at the time of Pharmacodynamic assessments | up to 10 hours post dosing
Plasma concentration of Oxycodone hydrochloride at the time of Pharmacodynamic assessments | up to 10 hours post dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational center, City Name, United Kingdom